CLINICAL TRIAL: NCT03939221
Title: Measure the Meridian Energy Change of Terminal Hospice Patient Via Meridian Energy Analysis Device to Evaluated the Relationship of Clinical Symptoms and Alternative Medicine Effect.
Brief Title: Measure the Meridian Energy Change of Terminal Hospice Patient Via Meridian Energy Analysis Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CCH-181018
Record Dates: First submitted 2019-04-07; First posted 2019-05-06 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2019-01

CONDITIONS: Hospice; Survival; Alternative Medicine; Skin Electric Conductance
Keywords: skin electric conductance; survival period; complementary and alternative medicine
MeSH Terms: interventions — Acupressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention of infrared lamp and acupressure (Experimental): Measure the ankle and wrist acupoints skin conductance to evaluate the basic condition of terminal hospice patients. Then investigators use the infrared lamp and acupressure(tender points, PC6(neiguan) and ST36(zusanli) for one minutes) for our patient for the cold limbs, pain control and constipation problems.
  Interventions: Behavioral: Infrared Lamp and Acupressure

INTERVENTIONS:
Behavioral: Infrared Lamp and Acupressure — Measure the ankle and wrist acupoints skin conductance to evaluate the basic condition of terminal hospice patients. Then investigators use the infrared lamp and acupressure(tender points, PC6 and ST36 for one minutes) for our patient for the cold limbs, pain control and constipation problems.

SUMMARY:
In the hospice ward, there are lots of suffered hospital patients with multiple physical discomfort related to terminal disease. Investigators want to use an objective measure instrument to monitor the effects of complementary and alternative medicine and clinical symptoms. First, investigators use the Meridian Energy Analysis Device (MEAD) to measure the bilateral 12 Yuan points (primary points) of terminal hospice patients. It provides the prediction value between terminal disease and the change of different meridian energy. Besides, the meridian energy value maybe predict the survival period. Then, the intervention of complementary and alternative medicine can also monitor via MEAD.

DETAILED DESCRIPTION:
In the hospice ward, there are lots of suffered hospital patients with multiple physical discomfort related to terminal disease. It may be caused by cancer or multiple kinds of organ failure. The terminal hospital patients have symptoms such as pain, dyspnea, fatigue, nausea, vomiting, poor appetite, constipation, ileus or edema…, etc. Investigators want to use an objective measure instrument to monitor the effects of complementary and alternative medicine.

First, investigators use the Meridian Energy Analysis Device (MEAD) to measure the bilateral 12 Yuan points (primary points) of terminal hospice patients (divided to cancer, multiple kinds of organ failure). It provides the prediction value between terminal disease and the change of different meridian energy. Besides, the meridian energy value maybe predict the survival period. Then, investigators use the intervention of complementary and alternative medicine (like infrared lamp and acupressure…, etc.) to improve the quality of life in the terminal hospice patients. Also, investigators will use the Meridian Energy Analysis Device, pain scale, vital signs and quality of life scale (SF-36) to evaluate the effects of complementary and alternative medicine.

ELIGIBILITY:
Inclusion Criteria:

* Patients lived at our Changhua Christian Hospital hospice ward
* From 2019-02~2020-12, age 20 to 99 years old, volunteer patient

Exclusion Criteria:

* Unwillingness
* Wound or amputation near wrist or ankle
* Severe agitation or seizure patients

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
The change of 24 points skin electric conductance over bilateral wrist and foot in terminal patients | through hospitalization period, an average of 1 month (after admission baseline evaluation and till discharge)
  Investigators use the meridian energy analysis device to measure the 24 points skin conductance over bilateral wrist and foot. The meridian energy analysis device is an electrophysiology tool to measure the skin micro-electrical currents(range from 0uA to 200uA). The higher skin conductance stands for better condition of patient. Investigators will evaluate the relationship between the skin conductances and clinical symptoms. Then investigators will check the effect via the skin electric conductance before and after the infrared lamp and acupressure intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Cheng Chung, Bachelor, Study Chair — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan